CLINICAL TRIAL: NCT02599883
Title: Impact of Low-dose Computed Tomography on the Management of Chronic Obstructive Pulmonary Disease Patients: an Evidence-based Study
Brief Title: Evidence-based Analysis of Low-dose CT in Management of COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Nicola Sverzellati, Professor, MD, PhD, Azienda Ospedaliero-Universitaria di Parma
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ImagingCOPD_Multicenter
Record Dates: First submitted 2015-11-04; First posted 2015-11-09 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Diagnostic Imaging; Disease Management; Clinical Decision Support Systems; Cost-Utility Analysis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MulticenterRecruitment (Experimental): COPD phenotypization by Low-Dose Computed Tomography
  Interventions: Radiation: Low-Dose Computed Tomography

INTERVENTIONS:
Radiation: Low-Dose Computed Tomography — Low-Dose Computed Tomography will be administered to COPD patients as part of COPD phenotypization.

SUMMARY:
Background: Chronic obstructive pulmonary disease (COPD) is the fourth leading cause of chronic morbidity and mortality worldwide. There is debate about diagnosis and management of COPD because it was described as complex syndrome accounting for various pulmonary and extrapulmonary abnormalities. As a result, there is consensus that both clinical evaluation and pulmonary function tests (PFTs) data by themselves do not adequately describe the complexity of the disease. The chest radiograph is the sole imaging examination recommended for the routine evaluation of these patients by the physicians guidelines (GOLD guidelines),which, however, are also debating on the utility of computed tomography (CT) in this setting. Indeed, a number of studies reported a dramatic increasing use of CT of the chest for COPD assessment, in both clinical and research settings. COPD assessment by CT seems to improve the accuracy and completeness of the clinical evaluation of these patients. Nevertheless, the clinical utility of CT has yet to be proved by prospective studies or defined by guidelines.

Objectives: To evaluate the change in the diagnosis and management of COPD when multiple CT-derived information is added to pre-test evaluation.

Methods: Four pulmonologists with various expertise in the field will review clinical data, PFTs results, and chest radiographs of 200 consecutive COPD patients diagnosed according to current guidelines. Therefore, after two months from the first evaluation, the pulmonologists will review the clinical and PFTs records with comprehensive information about low-dose CT (LDCT) previously performed in a week from the chest radiograph. Information about LDCT findings will include qualitative assessment by an experienced chest radiologist and quantitative analysis by means of an innovative 3D imaging dedicated software. Phenotype assessment and patient care decisions (e.g. therapeutic and follow-up strategies, need of additional tests etc.) will be recorded before and after assimilation of LDCT data.

Expected results: This evidence-based prospective study will test the impact of chest LDCT on management of COPD patient. In addition, the level of agreement between pulmonologists in terms of diagnosis and therapeutic strategies will be assessed. Furthermore, the study will evaluate the need for additional tests referable to LDCT information and their impact on the health care system (e.g. in terms of additional costs).

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis according to ATS/ERS criteria (post-bronchodilator FEV1 to FVC ratio < 0.7);
* clinical stability, namely no acute exacerbation in the previous 4 weeks;
* clinical indication for low-dose computed tomography (LDCT) to investigate bronchiectasis, interstitial lung disease, or pulmonary hypertension.

Exclusion Criteria:

* pregnancy;
* patients with congenital or acquired immune deficit;
* patients with lung transplantation;
* patients under oxygen therapy;
* patients with diagnosis of asthma or other clinically relevant pulmonary disease other than COPD.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Impact of diagnostic imaging in assessing COPD by qualitative and quantitative evaluation (questionnaire) | Up to 3 years
  To quantify the refinement of the diagnosis of COPD patients when LDCT data are added to standard evaluation, namely, conventional clinical-functional assessment and chest radiography.
Clinical management of COPD in relation to therapy adjustment (questionnaire) | Up to 3 years
  To describe the change in management of COPD patients when LDCT data are added to standard evaluation, namely, conventional clinical-functional assessment and chest radiography.

SECONDARY OUTCOMES:
Intra-observer agreement before and after disclosure of LDCT features (questionnaire) | Up to 3 years
  To assess the intra-observer agreement of pulmonologists before and after assimilation of LDCT data.
Inter-observer agreement (questionnaire) | Up to 3 years
  To assess changes in inter-observer agreement between pulmonologist before and after assimilation of LDCT data.
Additional costs derived from change in management of COPD after disclosure of LDCT features (comparison of costs) | Up to 3 years
  To evaluate additional costs for the regional health care system deemed by assimilation of LDCT data.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Sverzellati, MD, PhD, Principal Investigator — Università di Parma